CLINICAL TRIAL: NCT03647943
Title: Neuromodulation Augmented Cognitive Training to Improve Cognitive Flexibility in Anorexia Nervosa
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: COVID-19 pandemic (residential treatment center closed to visitors)
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: PSYCH-2018-26509
Record Dates: First submitted 2018-07-24; First posted 2018-08-27 (Actual); Last update posted 2022-03-14 (Actual); Status verified 2022-02

CONDITIONS: Active tDCS; Sham tDCS
MeSH Terms: interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: One arm of this study is a sham condition; both tDCS and sham tDCS conditions are blinded to participants and study assessor/s.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active tDCS (Experimental): Participants will receive 10 sessions of active tDCS + cognitive training.
  Interventions: Device: Transcranial direct current stimulation
- Sham tDCS (Sham Comparator): Participants will receive 10 sessions of sham tDCS + cognitive training.
  Interventions: Device: Sham transcranial direct current stimulation

INTERVENTIONS:
Device: Transcranial direct current stimulation — Transcranial direct current stimulation, involving low-levels of electrical stimulation applied to the right and left DLPFC will be used in conjunction with cognitive training for 46 minutes.
  Arms: Active tDCS
Device: Sham transcranial direct current stimulation — Sham transcranial direct current stimulation, involving no electrical stimulation will be used in conjunction with cognitive training for 46 minutes.
  Arms: Sham tDCS

SUMMARY:
The purpose of the study is to evaluate the use of a new brain stimulation tool called transcranial direct current stimulation (tDCS). tDCS is a new technique used to stimulate the brain. The investigators believe that it may help to change brain function in individuals with anorexia nervosa. The brain stimulation occurs outside the head. The tDCS procedure involves applying a small amount of electrical current across the scalp, for a short period of time. This small electrical current is able to change the electrical activity inside areas of the brain. In the current study, the investigators will ask participants to complete computer-based brain training sessions. While participants do the brain training exercises, they will receive either real tDCS for "sham" tDCS. "Sham" tDCS means that participants might feel sensations like tingling or vibrations from the tDCS machine, but will not actually receive the electrical current. Investigators will also ask participants to complete several tests to assess changes in brain function. The information gained from this study will help investigators to understand how tDCS could be used to improve brain function and learning in individuals with anorexia nervosa.

ELIGIBILITY:
Inclusion Criteria:

* Age 18+ years
* Documented enrollment in residential-level treatment at The Emily Program and meeting criteria for AN (BMI <18.5).
* Participant must be capable of giving informed consent, based on University of California San Diego (UCSD) Brief Assessment of Capacity to Consent (UBACC)39 risk assessment, which has been uploaded to ETHOS.
* Sufficient spoken English so as to be able to comprehend testing procedures.

Exclusion Criteria:

* Substance abuse in the participant
* Neurological condition or other developmental disorder
* Serious psychiatric disorder known to affect brain functioning and cognitive performance
* Medical instability, which will be evident based on required admittance status in the residential treatment facility from which participants will be recruited. (The Emily Program residential treatment patients are followed closely by a medical provider, who routinely assesses medical stability throughout the duration of each patient's stay in the treatment facility; therefore, if a participant is not currently a patient in this setting and/or has been recently discharged from residential treatment setting due to medical need to receive higher level of care/inpatient-level care, they will be excluded from enrollment in this study).
* MRI contraindication [based on Center for Magnetic Resonance Research (CMRR) prescreening protocol]
* tDCS contraindication (e.g., history of craniotomy, history of metallic cranial plates, screws, implanted devices).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-08-30 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Number of participants with treatment-related adverse events as assessed by CTCAE v4.0 and rate of treatment dropout in treatment-seeking adults with AN receiving treatment in a residential treatment program for eating disorders. | Through study completion, an average of 1 year.
  Treatment-related adverse events will be assessed by CTCAE v4.0 criteria. Participant dropout will be examined in effort to evaluate whether individuals with AN will tolerate the procedures and remain in the study. This will be evinced by less than 20% dropout over the course of active tDCS and cognitive training.
Change from Baseline to End of Treatment Set-Shifting Task Performance Following 10-session tDCS + Cognitive Training Intervention Protocol. | Through study completion, an average of 1 year.
  Changes in cognitive flexibility will be assessed by examining differences between baseline and end of treatment performance on reversal learning task.
Change from Baseline to End of Treatment Resting State and Task-based Functional Magnetic Resonance Imaging (fMRI) Activation during Reversal Learning Task Following 10-session tDCS + Cognitive Training Intervention Protocol. | Through study completion, an average of 1 year.
  Changes in brain circuitry assessed during resting state and task-based fMRI will be assessed to examine whether active tDCS is associated with greater change in associated circuitry, as compared with sham tDCS.

SECONDARY OUTCOMES:
Change in Eating Disorder Examination (EDE) Scores from Baseline to End of Treatment | Through study completion, an average of 1 year.
  Change in eating disorder psychopathology, measured by the EDE, will be evaluated over the course of a 10-session tDCS + cognitive training intervention to determine whether tDCS is associated with significant change in eating pathology among individuals with Anorexia Nervosa.

CONTACTS AND LOCATIONS:
Overall Officials: Kelvin O Lim, MD, PhD, Principal Investigator — University of Minnesota
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No
There is no plan to share Individual Participant Data (IPD) with other researchers.